CLINICAL TRIAL: NCT00402194
Title: Treating the Endothelium to Restore Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IU-IRB-0301-08
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Insulin Resistance; Impaired Glucose Tolerance; Pre-diabetes
Keywords: Obesity; Insulin resistance; Impaired glucose tolerance; pre-diabetes
MeSH Terms: conditions — Obesity; Insulin Resistance; Glucose Intolerance | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Losartan — Tablet, 100mg, once per day for 3 months

SUMMARY:
A study of 12 weeks' treatment with losartan or placebo, to test the hypothesis that RAS inhibition will improve insulin' vascular actions and therefore improve insulin sensitivity in skeletal muscle.

DETAILED DESCRIPTION:
Recent studies suggesting an effect of cardiovascular therapies to prevent diabetes remain unexplained. We hypothesize that these therapies improve vascular endothelial function allowing improved actions of insulin in the vasculature, which comprise a significant portion of insulin's metabolic action. We therefore propose to measure insulin-mediated glucose disposal and insulin-mediated vasodilation before and after 12 weeks' therapy with Losartan (an angiotensin receptor blocker) or placebo, in a randomized design. Subjects will include 28 subjects with impaired glucose tolerance, which is generally accompanied by both insulin resistance and impaired vascular function. With this number of participants we have a 90% chance of showing a statistically significant and clinically meaningful effect of insulin on leg vascular resistance, and an even higher chance of showing a difference in insulin's metabolic effects. Exclusion criteria will include frank hypertension, diabetes, or hypercholesterolemia, and biochemical or other contraindications to losartan therapy. The primary endpoint for statistical analysis will be the invasive measure of insulin-stimulated endothelial function. We anticipate an improvement in both vascular and metabolic measures of insulin action following Losartan therapy but no change from untreated baseline following placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 20-55
* Male and female
* Obese, defined as Males: BMI >28 or > 30% fat by DEXA scan or Bod Pod; Females: BMI >30 or > 33% fat by DEXA scan or Bod Pod
* Weight stable over at least 4 months

Exclusion Criteria:

* Diabetes mellitus (ADA criteria)
* Age <20 or > 55 yrs
* Blood pressure >160/90 or < 90/65 mmHg
* Total cholesterol >240 or LDL cholesterol >160 mg/dL
* Baseline elevations in AST or ALT > 3X ULN
* Baseline elevation in creatinine >1.6 ng/mL
* Unexplained baseline elevation in creatine kinase > 3X ULN
* Concurrent significant chronic medical illness including, but not limited to, human immunodeficiency virus infection, Syphilis, hepatitis B infection, or hepatitis C infection
* Pregnancy
* Known hypersensitivity or intolerance to the study agents

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-06; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital GCRC, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by word of mouth and flyers posted in key locations on campus.
Groups:
- Treatment: Treatment with 100mg of losartan daily. Outcomes measured before and after 3 months of treatment.
- Placebo: Treatment with double blinded placebo daily. Outcomes measured before and after 3 months of treatment.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Treatment with 100mg of losartan daily or placebo. Outcomes measured before and after 3 months of treatment.
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (8.7) | 36.5 (10.1) | 38.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Leg Blood Flow Response to Insulin
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 9 | 8
Liters/minute
  Baseline Leg Blood Flow | 0.24 (0.05) | 0.26 (0.05)
  Insulin stimulated leg blood flow | 0.353 (0.327) | 0.046 (0.049)

2. Primary Outcome: Insulin-stimulated Leg Glucose Uptake
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmol/min
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 9 | 8
mmol/min | 0.42 (0.08) | 0.30 (0.09)

ADVERSE EVENTS:
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No